CLINICAL TRIAL: NCT01757119
Title: Study of the Pharmacokinetics of Serum Iron After Single Oral Administration of Ferrous Sulphate Supplement in Women With Iron Deficiency Anaemia
Brief Title: Ferrous Sulphate Supplement in Women With Iron Deficiency Anaemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L00008 CP 1 01; 2012-002190-63 (EudraCT Number)
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate, mucin drug combination

ARMS (1):
- Drug (Experimental)
  Interventions: Drug: Tardyferon 80 mg

INTERVENTIONS:
Drug: Tardyferon 80 mg — Oral administration (2 tablets)

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of serum iron (the amount of iron in blood) after single oral administration of 2 tablets of L0008 80 mg (as ferrous sulphate) in women with iron deficiency anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years old with iron deficiency anaemia
* haemoglobin level between 85 g/L and 105 g/L
* serum ferritin level < 15 µg/L
* D14 + 7 days of the menstruation cycle on the day of pharmacokinetic evaluation
* Standard diet

Exclusion Criteria:

* - Anaemia related to other causes than iron deficiency and particularly inflammatory anaemia, anaemia due to marrow failure, haemopathy, haemoglobinopathies (sickle cell disease, thalassemia), haemolytic anaemia, anaemia due to acute haemorrhage, or anaemia related to chronic renal failure,
* Haemochromatosis or iron overload of secondary origin (blood transfusion),
* Long term treatment known to modify iron absorption,
* Gastro duodenal ulcer,
* Inflammatory bowel disease or any digestive disease which could modify iron absorption,
* Fructose intolerance, syndrome of malabsorption of glucose, galactose, deficit of sucrase-isomaltase,
* Serious or progressive disease (cardiac, pulmonary, hepatic, renal, haematological, malignancy, autoimmune disease, infectious disease or neuropsychiatric disorders),
* Surgery undergone within 1 month prior to selection visit or a surgery planned during the study realization.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of serum iron after single oral administration of ferrous sulphate supplement | Up to 24 hours
  Pharmacokinetic profile of serum iron after single oral administration of ferrous sulphate supplement by measuring Maximum Plasma concentration, Time of Maximum Concentration, Area under the iron plasma concentration curve.

SECONDARY OUTCOMES:
Tolerability of single administration (reported adverse events) | Up to 24 hours
  Tolerability by evaluating the number of subjects with emergent adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - Iași
  - Timișoara